CLINICAL TRIAL: NCT04267068
Title: Single Session Intervention to Prevent Common Mental Disorders and Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 1219218
Record Dates: First submitted 2019-11-05; First posted 2020-02-12 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Online growth mindset interactive article followed by equal length interactive article describing the relationship between modifiable risk factors (MRF) and mental health outcomes
  Interventions: Behavioral: Growth Mindset and Modifiable Risk Factor Information
- Control (Active Comparator): Online daily activity scheduling interactive article (control)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Growth Mindset and Modifiable Risk Factor Information — 15 minute interactive article describing neuroplasticity followed by 15 minute interactive article describing modifiable risk factors for depression and anxiety
  Arms: Intervention
Behavioral: Control — 30 minute interactive article describing symptoms of depression and anxiety, common concerns of college student
  Arms: Control

SUMMARY:
The present study aims to determine the effect of presenting psychoeducation emphasizing "growth-mindset," and information on depression and anxiety symptom severity. The investigators hypothesize that psychoeducation emphasizing that mental health is malleable will increase the participant's engagement with risk factors outlined in the intervention

DETAILED DESCRIPTION:
Depression and anxiety disorders (or common mental disorders; CMDs) are increasingly common among college students, with rates comparable to the general population. As such, brief, scalable and transdiagnostic prevention efforts targeting CMDs are needed. In order to address this need, this study aims to evaluate the impact of a single session intervention (SSI) utilizing growth mindset (GM) on CMD symptom severity and investigate the mediating role of changes in modifiable risk factors in the relationship between intervention and CMD symptom reduction. The intervention will adapt existing GM interventions for college students to engage mechanisms in the prevention and management of common mental disorders including engagement in modifiable risk factors. College students will be randomly assigned to complete either a GM intervention or a psychoeducation control.

ELIGIBILITY:
Inclusion Criteria:

* Age 17-26
* College student at the University of Nevada, Reno

Exclusion Criteria:

* Under the age of 17, over the age of 26
* Participated in pilot study
* Not a college student at the University of Nevada, Reno

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 375 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer & Williams, 2001) | 6 months
  9-item questionnaire associated containing one item for each symptom of MDD as specified by the DSM. Items consist of a 4-point Likert scale (0="Not at all" to 3="Nearly every day"). Minimum score is 0, maximum score is 27. Higher scores indicate greater depression severity.
Generalized Anxiety Disorder-7 (GAD-7; Spitzer, Kroenke, Williams & Lowe, 2006) | 6 months
  7-item scale, common, brief measure of anxiety symptom severity. Items consist of a 4-point Likert scale (0="Not at all" to 3="Nearly every day"). Minimum score is 0, maximum score is 21. Higher scores indicate greater anxiety symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Papa, Ph.D., Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No